CLINICAL TRIAL: NCT01393626
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Centre Study To Investigate The Safety And Efficacy Of CP-690,550 For Induction Therapy In Subjects With Moderate To Severe Crohn's Disease
Brief Title: A Study To Investigate Safety And Efficacy Of CP-690,550 For Induction Therapy In Subjects With Moderate To Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921083; 2011-001733-16 (EudraCT Number)
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo
- 5mg BID (Experimental)
  Interventions: Drug: CP-690,550
- 10mg BID (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Placebo — oral tablets twice daily
  Arms: Placebo BID
Drug: CP-690,550 — oral tablets twice daily
  Arms: 5mg BID
Drug: CP-690,550 — oral tablets twice daily
  Arms: 10mg BID

SUMMARY:
This study investigates safety and efficacy of CP-690,550 in adult patients with moderate to severe Crohn's disease. The study hypothesis is that at least one dose of the tested drug is more effective than placebo (inactive drug).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 75 years at screening (upper age limit will be 64 years in India and 65 years in the Netherlands).
* Subjects with clinical diagnosis of Crohn's disease for at least 6 months prior to screening.
* Subjects with active moderate to severe ileal, ileocolic, or colonic CD defined by a baseline score of Crohn's Disease Activity Index (CDAI) of 220 to 450 at baseline.

Exclusion Criteria:

* Diagnosis of indeterminate colitis, ulcerative colitis (UC), or clinical findings suggestive of UC.
* Subjects diagnosed with Crohn's disease but without previous exposure to treatment (i.e., treatment-naïve).
* Subjects receiving the following treatment for Crohn's disease:
* Azathioprine, 6-mercaptopurine or methotrexate within 2 weeks prior to baseline.
* Anti-TNFα therapy within 8 weeks prior to baseline.
* Interferon therapy within 8 weeks prior to baseline.
* Cyclosporine, mycophenolate, or tacrolimus within 4 weeks prior to baseline.
* Intravenous corticosteroids within 2 weeks prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (139):
- United States (72):
  - ACRI - Phase 1, LLC, Anaheim, California
  - Advanced Clinical Research Institute - Phase 1, LLC, Anaheim, California
  - AGMG Endoscopy Center, Anaheim, California
  - Alliance Clinical Research, Oceanside, California
  - Alliance Clinical Research, LLC, Poway, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Clinical Research Of The Rockies, Lafayette, Colorado
  - Endoscopy Center of the Rockies - Longmont, Longmont, Colorado
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Metropolitan Gastroenterology Group, PC, Washington D.C., District of Columbia
  - Gasteroenterology Consultants of Clearwater, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Citrus Surgery & Endoscopy Center (Colonoscopy & Biopsy Only), Crystal River, Florida
  - Shands Endoscopy Center, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Investigational Drug Service, Gainesville, Florida
  - Shands Medical Plaza and Cancer Center, Gainesville, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center (Colonoscopy Only), Inverness, Florida
  - FQL Research, LLC, Miramar, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gulfshore Endoscopy Center (Endoscopies Only), Naples, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Heartland Medical Research, Inc (Administrative Only), Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - Iowa Endoscopy Center (Colonoscopy Only), Clive, Iowa
  - Iowa Radiology (MRI, X-Ray Only), Clive, Iowa
  - Cotton-O'Neil Clinical (X-Ray), Topeka, Kansas
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Stormont-Vail MRI Center of Kansas, Topeka, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - Metropolitan Gastroenterology Group, PC, Chevy Chase, Maryland
  - East Ann Arbor Health and Geriatrics Center, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Charlotte Radiology (Chest X-Ray Only), Charlotte, North Carolina
  - University Hospitals Chagrin Highlands Health Center, Beachwood, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Gastroenterology, Inc., Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - University Hospitals Westlake Medical Center, Westlake, Ohio
  - Great Lakes Gastroenterology, Willoughby, Ohio
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - UT Health Science Center, Houston, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Cardiology Consultants (ECG Site Only), Norfolk, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - MRI & CT Diagnostics, Virginia Beach, Virginia
  - The Center for Digestive Health, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research - GI Associates, LLC, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Medical Diagnostic Imaging (MDI) X-ray and MRI only, Milwaukee, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
  - GI Associates, Wauwatosa, Wisconsin
- Australia (3):
  - Nepean Public Hospital, Kingswood, New South Wales
  - Monash Medical Center, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Bulgaria (4):
  - 4-MBAL, Parvo vatreshno otdelenie, Sofia
  - MBAL Sveti Ivan Rilski, Klinika po Gastroenterologia, Sofia
  - MBAL Voennomeditsinska Akademia, Sofia
  - MBAL Sofiamed OOD, Otdelenie po gastroenterologia, Sofia
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - Office of Dr. David C. Pearson, Victoria, British Columbia
  - Office of Drs. Ranjith Andrew Singh and Jamie D. Papp, Victoria, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Inflammatory Bowel Disease Centre, Montreal General Hospital, McGill University Health Centre, Montreal, Quebec
- Croatia (2):
  - University Hospital Centre Rijeka, Rijeka
  - University Hospital Center Zagreb, Zagreb
- Czechia (3):
  - Medial Pharma spol.s.r.o., Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - RDG centrum s.r.o., Hradec Králové
- France (3):
  - Hopital Huriez, CHRU de Lille, Lille
  - Hopital Haut-Leveque, Pessac
  - Hopital Robert Debre, Reims
- Germany (5):
  - Charite - Campus Berlin Mitte, Berlin
  - Charite Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Universitaetsklinikum Ulm, Klinik fuer Innere Medizin I, Ulm
- General Hospital of Athens "Evangelismos",1st Gastroenterology Department, Kolonaki Athens, Greece
- Hungary (8):
  - Magyar Honvedseg Honvedkorhaz II. telephely/Gasztroenterologiai Osztaly, Budapest
  - Peterfy Sandor Utcai Korhaz, Rendelointezet es Baleseti Kozpont, I. sz. Belgyogyaszat, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak/I. Belgyogyaszat es Gastroenterologia, Budapest
  - Pannonia Maganorvosi Centrum Kft, Budapest
  - Laboratorium Kft. Fovarosi es Pest Megyei Mikrobiologiai Laboratorium, Budapest
  - Bugat Pal Korhaz Egeszsegugyi Szolgaltato Kozhasznu Nonprofit Kft, Gyöngyös
  - Somogy megyei Kaposi Mor Oktato Korhaz / Belgyogyaszati osztaly, Kaposvár
  - Clinfan Kft., Szekszárd
- Israel (4):
  - Digestive Diseases Institute, Shaare Zedek Medical Center, Jerusalem
  - Dept. of Gastroenterology & Hepatology, Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (8):
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Toho University Sakura Medical Center, Chiba
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
- South Africa (2):
  - Kingsbury Hospital, Cape Town, Western Cape
  - Parklands Medical Centre, Durban
- South Korea (3):
  - Severance Hospital, Yeonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - ASAN Medical Center, Seoul
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
- Ukraine (6):
  - State Institution "Institute of Gastroenterology of AMS of Ukraine", Dnipropetrovsk
  - Donetsk National Medical University n.a M. Gorky, Faculty of Internal Medicine #2,, Donetsk
  - State Institution "Institute of Therapy n.a. L.T. Mala of AMS of Ukraine", Kharkiv
  - Lviv National Medical University n.a Danylo Halytsky, Faculty of Surgery#1 with Proctology Course, Lviv
  - Municipal Institution "Odesa Regional Clinical Hospital". Odesa Regional Centre of Gastroenterology., Odesa
  - Medical Clinical Research Center Health Clinic on base LLC "Medical Diagnostic Center Slaomed", Vinnitsa

REFERENCES:
- [Derived] Panes J, Sandborn WJ, Schreiber S, Sands BE, Vermeire S, D'Haens G, Panaccione R, Higgins PDR, Colombel JF, Feagan BG, Chan G, Moscariello M, Wang W, Niezychowski W, Marren A, Healey P, Maller E. Tofacitinib for induction and maintenance therapy of Crohn's disease: results of two phase IIb randomised placebo-controlled trials. Gut. 2017 Jun;66(6):1049-1059. doi: 10.1136/gutjnl-2016-312735. Epub 2017 Feb 16. PMID 28209624
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921083&StudyName=A%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%2C%20Parallel%20Group%2C%20Multi-centre%20Study%20To%20Investigate%20The%20Safety%20And%20Efficacy%20Of%20Cp-690%2C550%20For%20Induction%20Therapy%20In%20Subjects%20With%20Moderate%20To%20Severe%20Crohn%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 280 participants were randomized to treatment but only 279 participants received treated.
Groups:
- Placebo: Placebo tablets to match tofacitinib 5 milligrams (mg) for oral administration twice daily (BID) for 8 weeks.
- Tofacitinib 5 mg BID: Tofacitinib tablets for oral administration at a dose of 5 mg BID for 8 weeks.
- Tofacitinib 10 mg BID: Tofacitinib tablets for oral administration at a dose of 10 mg BID for 8 weeks.
- Tofacitinib 15 mg BID: Tofacitinib tablets for oral administration at a dose of 15 mg BID for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Started | 91 | 86 | 86 | 16
Completed | 73 | 74 | 74 | 15
Not Completed | 18 | 12 | 12 | 1
Not completed — Adverse Event | 2 | 1 | 5 | 0
Not completed — Did not meet entrance criteria | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 6 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set - included all participants who received at least one dose of study medication.
Groups:
- Placebo: Placebo tablets to match tofacitinib 5 mg for oral administration BID for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Total
Number analyzed (Participants) | 91 | 86 | 86 | 16 | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (11.7) | 40.2 (11.5) | 39.3 (13.7) | 41.3 (14.3) | 39.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 32 | 47 | 7 | 146
  Male | 31 | 54 | 39 | 9 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission (as Defined by a Crohn's Disease Activity Index [CDAI] Score of Less Than [<] 150 Points) at Week 8
Description: Clinical remission was a CDAI < 150 points. CDAI is a composite index consisting of a weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's diary kept while on study. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Week 8
Population: Full analysis set (FAS) - included all randomized participants who received at least 1 dose of investigational product and who had a qualified CDAI score calculated using the hematocrit value measured at baseline visit (Day 1). Participants with missing values were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
Percentage of Participants | 36.67 [26.75 to 47.49] | 43.53 [32.80 to 54.72] | 43.02 [32.39 to 54.15]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Tofacitinib-Placebo; Test type: Superiority or Other; p = 0.3249, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.86, 95% CI 2-sided [-7.64 to 21.36]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 10 mg BID; Tofacitinib-Placebo; Test type: Superiority or Other; p = 0.3916, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.36, 95% CI 2-sided [-8.09 to 20.80]

2. Secondary Outcome: Percentage of Participants in Clinical Remission (CDAI <150) at Weeks 2 and 4
Description: Clinical remission was a CDAI <150 points. CDAI is a composite index consisting of a weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's diary kept while on study. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Weeks 2 and 4
Population: FAS, participants with missing values were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
Percentage of Participants
  Week 2 | 10.00 [4.68 to 18.14] | 9.41 [4.15 to 17.71] | 9.30 [4.10 to 17.51]
  Week 4 | 21.11 [13.21 to 30.99] | 24.71 [15.99 to 35.25] | 22.09 [13.86 to 32.33]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response-70 (as Defined by a Decrease in CDAI Score of at Least 70 Points From Baseline) at Weeks 2, 4, and 8
Description: Clinical response-70 was defined as a reduction in CDAI score from baseline of at least 70 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: FAS, participants with missing values were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
Percentage of Participants
  Week 2 | 37.78 [27.77 to 48.62] | 47.06 [36.13 to 58.19] | 44.19 [33.48 to 55.30]
  Week 4 | 50.00 [39.27 to 60.73] | 57.65 [46.45 to 68.30] | 56.98 [45.85 to 67.61]
  Week 8 | 62.22 [51.38 to 72.23] | 76.47 [66.03 to 85.00] | 74.42 [63.87 to 83.22]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Response-100 (as Defined by a Decrease in CDAI Score of at Least 100 Points From Baseline) at Weeks 2, 4, and 8
Description: Clinical response-100 was defined as a reduction in CDAI score from baseline of at least 100 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: FAS, participants with missing values were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
Percentage of Participants
  Week 2 | 23.33 [15.06 to 33.43] | 34.12 [24.18 to 45.20] | 32.56 [22.84 to 43.52]
  Week 4 | 37.78 [27.77 to 48.62] | 48.24 [37.26 to 59.34] | 45.35 [34.58 to 56.45]
  Week 8 | 54.44 [43.60 to 64.98] | 70.59 [59.71 to 79.98] | 68.60 [57.70 to 78.19]

5. Secondary Outcome: Percentage of Participants Achieving Either Clinical Response-100 or Clinical Remission (CDAI<150) at Weeks 2, 4, and 8
Description: Clinical response-100 was defined as a reduction in CDAI score from baseline of at least 100 points. Clinical remission was a CDAI < 150 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: FAS, participants with missing values were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
Percentage of Participants
  Week 2 | 24.44 [16.00 to 34.64] | 34.12 [24.18 to 45.20] | 32.56 [22.84 to 43.52]
  Week 4 | 38.89 [28.79 to 49.74] | 49.41 [38.39 to 60.48] | 46.51 [35.68 to 57.59]
  Week 8 | 55.56 [44.70 to 66.04] | 71.76 [60.96 to 81.00] | 69.77 [58.92 to 79.21]

6. Secondary Outcome: CDAI Scores at Weeks 2, 4, and 8
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 2, 4, and 8
Population: FAS. Number of Participants Analyzed is the number of participants in the analysis set, n is the number of participants with non-missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
Score on a scale
  Week 2 (n=85, 78, 77, 16) | 258.04 (89.79) | 237.60 (67.87) | 241.21 (75.27) | 270.31 (90.78)
  Week 4 (n=81, 78, 71, 15) | 228.65 (102.01) | 213.38 (86.04) | 203.58 (86.69) | 228.27 (103.01)
  Week 8 (n=80, 77, 75, 15) | 194.90 (111.88) | 162.77 (87.67) | 159.08 (81.30) | 172.47 (119.28)

7. Secondary Outcome: C-Reactive Protein (CRP) Serum Concentrations at Weeks 2, 4, and 8
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
Milligrams per liter (mg/L)
  Week 2 (n=89, 84, 81, 16) | 17.28 (23.07) | 8.26 (11.40) | 8.56 (14.03) | 7.89 (9.42)
  Week 4 (n=83, 82, 78, 16) | 18.94 (31.26) | 8.17 (10.60) | 9.48 (21.35) | 10.33 (16.80)
  Week 8 (n=80, 77, 74, 15) | 18.12 (26.42) | 9.49 (15.33) | 6.55 (11.00) | 5.77 (7.74)

8. Secondary Outcome: Calprotectin Fecal Concentrations at Weeks 2, 4, and 8
Description: Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg per kilogram (mg/kg)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
mg per kilogram (mg/kg)
  Week 2 (n=81, 76, 73, 16) | 492.95 (664.51) | 384.81 (342.90) | 403.35 (352.57) | 455.10 (461.87)
  Week 4 (n=81, 82, 71, 16) | 493.26 (682.81) | 467.09 (377.65) | 359.30 (306.88) | 338.11 (391.65)
  Week 8 (n=75, 66, 72, 14) | 428.45 (479.36) | 417.70 (336.75) | 385.66 (316.71) | 349.61 (365.37)

9. Secondary Outcome: Tofacitinib Plasma Concentrations From 0 to 2 Hours Post Dose on Day 1 and at Week 8/Early Termination (ET) Visit
Description: Plasma samples were collected from participants for the determination of tofacitinib concentrations. Only samples from tofacitinib-treated participants were subsequently analyzed. Plasma concentration data are summarized by nominal sample collection times specified in the protocol, and actual sample collection times may be different.
Time Frame: Pre-dose, 20 minutes, 40 minutes, 1 hour, and 2 to 3 hours post-dose on Day 1 and Week 8/ET visit
Population: Pharmacokinetic analysis set - included all participants who received at least one dose of study medication and had at least one measurable plasma concentration. n is the number of observations (i.e. non-missing concentrations) at each timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 85 | 86 | 16
nanograms per milliliter
  Day 1, 0 hours (n=83, 83, 16) | 0.006687 (0.049144) | 1.193 (9.0312) | NA (NA) — Number of observations above the lower limit of quantification equals (=) 0.
  Day 1, 20 minutes (n=82, 83, 16) | 27.44 (27.335) | 62.28 (60.795) | 65.83 (63.232)
  Day 1, 40 minutes (n=82, 81, 16) | 41.03 (24.210) | 84.61 (47.470) | 151.4 (61.288)
  Day 1, 1 hour (n=83, 83, 16) | 41.22 (18.432) | 82.48 (40.782) | 149.9 (42.220)
  Day 1, 2 hours (n=83, 82, 16) | 31.85 (12.442) | 70.01 (24.838) | 106.1 (26.661)
  Week 8/ET, 0 hours (n=78, 72, 13) | 4.216 (7.1089) | 11.57 (21.453) | 23.89 (45.837)
  Week 8/ET, 20 minutes (n=70, 70, 12) | 25.89 (21.485) | 71.14 (54.969) | 127.6 (89.861)
  Week 8/ET, 40 minutes (n=70, 69, 12) | 37.75 (23.891) | 93.09 (46.471) | 148.7 (58.948)
  Week 8/ET, 1 hour (n=70, 69, 12) | 37.47 (21.384) | 83.14 (35.100) | 144.7 (48.137)
  Week 8/ET, 2 hours (n=72, 70, 13) | 27.61 (15.742) | 62.38 (27.505) | 92.03 (27.806)

10. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score and Domain Scores (Bowel Function, Emotional Status, Systemic Symptoms, and Social Function) at Baseline and Week 8/ET Visit
Description: The IBDQ is a psychometrically validated patient reported outcome (PRO) instrument for measuring disease-specific quality of life (QOL) in participants with inflammatory bowel disease (IBD). IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items are grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: bowel symptoms 10 to 70; systemic symptoms 5 to 35; emotional function 12 to 84; social function 5 to 35. For each domain, a higher score indicates better QOL. Total score is the sum of each item score, and ranged from 32 to 224 with a higher score indicating a better QOL. Positive change in total score indicated improvement in QOL.
Time Frame: Baseline, Week 8/ET visit
Population: FAS. N is the number of subjects in the analysis set, Number of Participants Analyzed is the number of subjects with non-missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Placebo: Placebo tablets to match tofacitinib 5 mg for oral administration BID for 8 weeks (N=90).
- Tofacitinib 5 mg BID: Tofacitinib tablets for oral administration at a dose of 5 mg BID for 8 weeks (N=85).
- Tofacitinib 10 mg BID: Tofacitinib tablets for oral administration at a dose of 10 mg BID for 8 weeks (N=86).
- Tofacitinib 15 mg BID: Tofacitinib tablets for oral administration at a dose of 15 mg BID for 8 weeks (N=16).
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 88 | 84 | 81 | 16
Score on a scale
  IBDQ Total Score, Baseline | 118.50 (28.48) | 117.89 (27.98) | 113.67 (28.45) | 124.19 (26.97)
  IBDQ Total Score, Week 8/ET | 144.99 (37.97) | 159.14 (35.39) | 156.64 (36.66) | 159.00 (47.98)
  Bowel Function Score, Baseline | 37.78 (8.17) | 37.39 (9.37) | 36.29 (7.72) | 37.50 (9.78)
  Bowel Function Score, Week 8/ET | 45.76 (12.19) | 50.94 (11.02) | 50.69 (11.02) | 52.50 (13.81)
  Emotional Status Score, Baseline | 45.88 (13.04) | 45.34 (13.27) | 44.55 (13.27) | 47.25 (10.41)
  Emotional Status Score, Week 8/ET | 56.31 (14.39) | 59.54 (13.78) | 58.32 (14.71) | 57.25 (20.07)
  Systemic Symptoms Score, Baseline | 15.22 (5.24) | 15.58 (4.36) | 14.60 (4.78) | 16.44 (5.35)
  Systemic Symptoms Score, Week 8/ET | 19.70 (6.51) | 22.24 (6.30) | 21.80 (6.27) | 22.88 (7.05)
  Social Function Score, Baseline | 19.62 (7.28) | 19.48 (6.62) | 18.23 (7.09) | 23.00 (6.29)
  Social Function Score, Week 8/ET | 23.23 (8.47) | 26.43 (7.57) | 25.83 (7.80) | 26.38 (9.58)

11. Secondary Outcome: Change From Baseline IBDQ Total Score and Domain Scores (Bowel Function, Emotional Status, Systemic Symptoms, and Social Function) at Week 8/ET Visit Using Analysis of Covariance (ANCOVA)
Description: IBDQ is a validated PRO instrument for measuring QOL in IBD consisting of 32 items scored from 1 (worst response) to 7 (best response). 32 items are grouped into 4 domains scored as follows: bowel symptoms 10 - 70; systemic symptoms 5 - 35; emotional function 12 - 84; social function 5 - 35. For each domain, higher score indicates better QOL. Total score is the sum of each item score, & ranged from 32 to 224 with a higher score indicating better QOL. Positive change in total score indicated improvement in QOL.
  Adjusted means were derived from an ANCOVA model with baseline value as covariate, treatment group & prior use of anti-tumor necrosis factor (TNF) alpha (α) treatments as factors.
  The 15 mg BID treatment group was closed to further enrolment early in the study by Protocol Amendment 5 after only 16 participants were enrolled in this group. Therefore, the efficacy analysis was not performed for this group as the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Week 8/ET visit
Population: FAS. N is the number of subjects in the analysis set, Number of Participants Analyzed is the maximum number of subjects with non-missing data.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 88 | 84 | 81
Score on a scale
  IBDQ Total Score | 26.58 (3.76) | 41.20 (3.90) | 40.05 (3.90)
  Bowel Function Score | 8.36 (1.23) | 13.76 (1.28) | 13.88 (1.28)
  Emotional Status Score | 10.33 (1.37) | 13.87 (1.42) | 12.54 (1.43)
  Systemic Symptoms Score | 4.41 (0.66) | 6.70 (0.69) | 6.68 (0.69)
  Social Function Score | 3.68 (0.79) | 7.03 (0.82) | 6.95 (0.82)

12. Secondary Outcome: Percentage of Participants With an IBDQ Total Score of Greater Than or Equal to (≥) 170 at Week 8/ET Visit
Description: The IBDQ is a psychometrically validated PRO instrument for measuring disease-specific QOL in participants with IBD. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is the sum of each item score, and ranged from 32 to 224 with a higher score indicating a better QOL. Positive change in total score indicated improvement in QOL.
Time Frame: Week 8/ET visit
Population: FAS
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 88 | 84 | 81 | 16
Percentage of Participants | 26.1 | 45.2 | 43.2 | 43.8

13. Secondary Outcome: Percentage of Participants With ≥16 Point Increase From Baseline in IBDQ Total Score at Week 8/ET Visit
Description: as for outcome 12
Time Frame: Week 8/ET visit
Population: FAS. Number of Participants Analyzed is the number of participants in the analysis set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
Percentage of Participants | 61.4 | 75.0 | 76.5 | 75.0

14. Secondary Outcome: Percentage of Participants With a Response to the Patient-Reported Treatment Impact Assessment (PRTI) at Week 8/ET Visit by Category
Description: The IBD Patient Reported Treatment Impact Modified (PRTI) questionnaire comprises 3 individual questions administered to the participant: participant satisfaction with study treatment; participant preference for study drug over prior treatment (this question on participant preference for study drug is prefaced by a simple question of previous treatment/s for IBD received in order to place the preference question into context) and participant willingness to re-use the study treatment again. Each of these questions (except the question on previous treatment, which is informational only) is scored on a 5 point Likert scale. PSA = Patient Satisfaction Assessment; PPTA = Patient Previous Treatment Assessment; PPA = Patient Preference Assessment; PWA = Patient Willingness Assessment.
Time Frame: Week 8/ET visit
Population: FAS. Number of Participants Analyzed is the number of participants in the analysis set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
Percentage of Participants
  PSA: Extremely dissatisfied | 17.0 | 6.0 | 7.4 | 6.3
  PSA: Dissatisfied | 10.2 | 9.6 | 6.2 | 0
  PSA: Neither satisfied nor dissatisfied | 25.0 | 19.3 | 16.0 | 25.0
  PSA: Satisfied | 40.9 | 45.8 | 43.2 | 25.0
  PSA: Extremely satisfied | 6.8 | 19.3 | 27.2 | 43.8
  PPTA: Injectable prescription medicines | 42.0 | 39.5 | 22.2 | 37.5
  PPTA: Prescription medicines taken by mouth | 37.5 | 44.4 | 56.8 | 43.8
  PPTA: Surgery | 2.3 | 2.5 | 0 | 0
  PPTA:Prescription medicines and surgery | 5.7 | 7.4 | 8.6 | 6.3
  PPTA: No treatment | 12.5 | 6.2 | 12.3 | 12.5
  PPA: Definitely prefer the drug I am receiving now | 33.0 | 42.2 | 48.1 | 56.3
  PPA: Slight preference for drug I'm receiving now | 19.3 | 27.7 | 22.2 | 25.0
  PPA: I have no preference either way | 28.4 | 19.3 | 13.6 | 18.8
  PPA: Slight preference for previous treatment | 9.1 | 2.4 | 7.4 | 0
  PPA: No, I definitely prefer my previous treatment | 10.2 | 8.4 | 8.6 | 0
  PWA: Would definitely want to use same drug again | 44.3 | 53.0 | 61.7 | 50.0
  PWA: Might want to use the same drug again | 11.4 | 24.1 | 17.3 | 37.5
  PWA: I am not sure | 20.5 | 10.8 | 8.6 | 6.3
  PWA: Might not want to use same drug again | 6.8 | 2.4 | 4.9 | 0
  PWA: Definitely not want to use same drug again | 17.0 | 9.6 | 7.4 | 6.3

15. Secondary Outcome: Short Form 36 Health Survey (SF-36) Component and Domain Scores at Baseline and Week 8/ET Visit
Description: The component and domain scores were scored using the United States (US) 1998 general population norms. The resulting norm-based T scores for both the SF-36 version 2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. Higher scores indicate better health-related QOL.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 87 | 84 | 81 | 16
Score on a Scale
  Physical component score, Baseline | 37.12 (7.66) | 38.49 (6.78) | 35.28 (8.49) | 37.09 (9.14)
  Physical component score, Week 8/ET | 40.84 (9.23) | 45.23 (8.85) | 44.29 (9.41) | 47.01 (7.97)
  Mental Component Score, Baseline | 36.50 (12.26) | 34.85 (11.68) | 35.84 (10.68) | 39.26 (11.85)
  Mental Component Score, Week 8/ET | 42.46 (11.21) | 43.69 (12.15) | 43.65 (11.87) | 42.73 (16.37)
  Physical Functioning Domain, Baseline | 43.73 (8.93) | 43.56 (8.81) | 41.36 (10.03) | 42.66 (9.04)
  Physical Functioning Domain, Week 8/ET | 46.55 (8.93) | 49.68 (8.43) | 48.37 (8.78) | 49.57 (8.99)
  Role Physical Domain, Baseline | 35.34 (9.94) | 36.36 (9.71) | 32.57 (10.92) | 37.68 (12.43)
  Role Physical Domain, Week 8/ET | 39.92 (10.64) | 44.49 (11.52) | 42.84 (11.59) | 44.39 (13.18)
  Bodily Pain Domain, Baseline | 34.69 (8.79) | 35.22 (8.44) | 33.32 (8.25) | 34.98 (8.23)
  Bodily Pain Domain, Week 8/ET | 40.81 (10.43) | 44.68 (11.29) | 45.10 (10.41) | 47.61 (11.21)
  General Health Domain, Baseline | 30.58 (7.21) | 31.37 (7.15) | 29.56 (7.52) | 32.08 (12.42)
  General Health Domain, Week 8/ET | 34.36 (8.50) | 36.79 (8.53) | 37.19 (10.75) | 37.98 (13.51)
  Vitality Domain, Baseline | 35.06 (9.70) | 34.66 (7.86) | 35.80 (9.05) | 37.55 (11.88)
  Vitality Domain, Week 8/ET | 41.20 (11.45) | 45.22 (11.94) | 44.60 (12.53) | 48.77 (13.41)
  Social Functioning Domain, Baseline | 34.71 (11.83) | 35.53 (11.69) | 33.83 (11.36) | 35.90 (10.61)
  Social Functioning Domain, Week 8/ET | 40.02 (12.33) | 45.01 (11.79) | 43.46 (11.43) | 43.63 (14.94)
  Role Emotional Domain, Baseline | 38.45 (13.98) | 37.20 (12.96) | 35.34 (13.23) | 39.12 (14.02)
  Role Emotional Domain, Week 8/ET | 43.06 (12.43) | 44.77 (12.46) | 43.76 (11.94) | 42.90 (16.58)
  Mental Health Domain, Baseline | 37.60 (12.30) | 35.95 (11.38) | 36.98 (11.09) | 41.27 (10.27)
  Mental Health Domain, Week 8/ET | 43.75 (11.02) | 43.58 (11.67) | 44.76 (11.64) | 43.00 (15.96)

16. Secondary Outcome: Change From Baseline SF-36 Component and Domain Scores at Week 8/ET Visit Using ANCOVA
Description: The component and domain scores were scored using the US 1998 general population norms. The resulting norm-based T scores for both the SF-36 version 2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. Higher scores indicate better health-related QOL.
  Adjusted means were derived from the ANCOVA model with baseline value as a covariate, treatment group and prior use of anti-TNF alpha treatments as factors.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 87 | 84 | 81
Score on a Scale
  Physical component score | 3.72 (0.927) | 7.28 (0.967) | 8.07 (0.956)
  Mental Component Score | 6.47 (1.143) | 7.88 (1.178) | 7.13 (1.180)
  Physical Functioning Domain | 3.01 (0.850) | 6.14 (0.876) | 5.59 (0.876)
  Role Physical Domain | 5.02 (1.152) | 8.76 (1.191) | 8.95 (1.183)
  Bodily Pain Domain | 6.41 (1.132) | 9.94 (1.174) | 11.10 (1.171)
  General Health Domain | 3.62 (0.897) | 5.55 (0.937) | 7.03 (0.933)
  Vitality Domain | 5.55 (1.190) | 9.84 (1.225) | 8.05 (1.233)
  Social Functioning Domain | 5.25 (1.163) | 9.72 (1.206) | 8.66 (1.204)
  Role Emotional Domain | 5.59 (1.222) | 7.28 (1.257) | 7.14 (1.260)
  Mental Health Domain | 6.46 (1.100) | 7.05 (1.136) | 7.41 (1.134)

17. Secondary Outcome: EuroQoL 5 Dimensions Questionnaire (EQ-5D) Utility Scores at Baseline and Week 8/ET Visit
Description: EQ-5D is a participant rated questionnaire to assess health-related QoL in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range from -0.594 to 1.000; a higher score indicates a better health state.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
Score on a Scale
  Utility Score, Baseline | 0.56 (0.29) | 0.58 (0.26) | 0.49 (0.31) | 0.61 (0.24)
  Utility Score, Week 8/ET | 0.64 (0.27) | 0.71 (0.28) | 0.71 (0.27) | 0.77 (0.30)

18. Secondary Outcome: Change From Baseline EQ-5D Utility Scores at Week 8/ET Visit Using ANCOVA
Description: EQ-5D is a participant rated questionnaire to assess health-related QoL via a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain & discomfort, anxiety & depression; 1 = better health state (no problems); 3 = worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain. Score is transformed to a total score ranging from -0.594 to 1.000; higher score indicates better health state. Adjusted means were derived from the ANCOVA model with baseline value as a covariate, treatment group & prior use of anti-TNFα treatments as factors.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 84 | 84 | 80
Score on a Scale | 0.08 (0.029) | 0.14 (0.030) | 0.16 (0.030)

19. Secondary Outcome: EQ-5D Visual Analogue Scale (VAS) Scores at Baseline and Week 8/ET Visit
Description: EQ-5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeters (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Number analyzed (Participants) | 90 | 85 | 86 | 16
mm
  VAS Score, Baseline | 46.83 (18.63) | 49.51 (18.03) | 42.74 (18.04) | 52.06 (24.11)
  VAS Score, Week 8/ET | 58.32 (21.31) | 67.07 (19.39) | 65.77 (19.71) | 69.81 (21.11)

20. Secondary Outcome: Change From Baseline EQ-5D VAS Scores at Week 8/ET Visit Using ANCOVA
Description: EQ-5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeters (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
  Adjusted means were derived from the ANCOVA model with baseline value as a covariate, treatment group & prior use of anti-TNF alpha treatments as factors.
  The 15 mg BID treatment group was closed to further enrolment early on in the study by Protocol Amendment 5 after only 16 participants were enrolled into this group. Therefore, the efficacy analysis was not performed for this group because the results may be difficult to interpret due to the small sample size.
Time Frame: Baseline, Week 8/ET visit
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 90 | 85 | 86
mm | 11.97 (2.166) | 19.56 (2.252) | 20.62 (2.222)

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent through and including 28 calendar days after last administration of study treatment (i.e. 11 weeks). Non-SAEs were recorded from time of first dose of study treatment through last participant visit (i.e. 15 weeks).
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID
Serious Adverse Events (participants affected / at risk) | 3/91 | 3/86 | 10/86 | 0/16
Other Adverse Events (participants affected / at risk) | 43/91 | 37/86 | 42/86 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Tofacitinib 5 mg BID (N=86) | Tofacitinib 10 mg BID (N=86) | Tofacitinib 15 mg BID (N=16)
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=91) | Tofacitinib 5 mg BID (N=86) | Tofacitinib 10 mg BID (N=86) | Tofacitinib 15 mg BID (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 7 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 6 | 5 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 5 | 7 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 5 | 0
Asthenia (General disorders) | 2 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 3 | 3 | 0
Pyrexia (General disorders) | 3 | 2 | 5 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 3 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 6 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 1 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 2 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 0
Headache (Nervous system disorders) | 7 | 8 | 5 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1/60 | 0 | 1/47 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Flushing (Vascular disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The PI must remove any previously undisclosed Confidential Information (other than the Study results themselves) before public release.